CLINICAL TRIAL: NCT00032526
Title: Classical Conditioning to Treat Allergic Airway Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: NCRR-M01RR02558-0180
Record Dates: First submitted 2002-03-25; First posted 2002-03-26 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Allergic Airway Disease
MeSH Terms: interventions — Adrenal Cortex Hormones

INTERVENTIONS:
Drug: Corticosteroids
Behavioral: Classical conditioning to corticosteroid

SUMMARY:
Most clinicians who care for patients with inflammatory airway diseases such as allergic rhinitis and asthma are aware of the negative effects of certain sights, sounds and smells that can precipitate clinical exacerbations in certain susceptible patients. This is thought to be due to subconscious associations between these observable stimuli paired and actual exposure to allergens that induce clinical symptoms. The severity and duration of these symptoms are typically related to levels of anxiety and/or depression in affected patients. Classical conditioning of the immune response has been described in many animal and some human studies in association with administration of immunosuppressive drugs. In successfully conditioned individuals, subsequent exposure to the conditioning stimulus alone produces immunosuppressive changes similar to those caused by the drugs themselves. Since disease exacerbating conditioning appears to be prevalent in allergic patients, these conditions make an excellent human model for understanding the relationships between classical conditioning, psychological stress (particularly anxiety and depression) and immune regulation. Thus this proposal will seek to examine the hypothesis that antiinflammatory effects of pharmacotherapeutic agents can be classically conditioned and are clinically effective due to changes in immunoregulatory imbalances known to occur in patients with allergic airway diseases. The effectiveness of this therapeutic approach will be significantly affected by levels of psychological stress and individual suggestibility. This will be investigated with the following Specific Aims: (1). Determine the relative effectiveness of classical conditioning by a novel gustatory stimulus paired with immunosuppressive doses of corticosteroid on in vivo and in vitro immune responses (allergen - specific vs. general) of patients before, during and after classical conditioning correlated with level of clinical response; (2) Determine the role of neuroendocrine mechanisms (particularly catecholamines) on the inducibility and duration of the conditioned immune responses; and (3) Investigate the influence of psychological stress levels (including anxiety and depression) and/or suggestibility on baseline immune changes, success and duration of the classical conditioning.

These data will help define parameters for classical conditioning in humans, establish a model to investigate mechanisms and serve as the basis for development of future interventional protocols for severe inflammatory diseases involving classical conditioning.

ELIGIBILITY:
Current history of allergic airway disease confirmed by positive skin tests. Included will be only those who have never tasted licorice or do not like the taste of licorice.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical School, Houston, Texas, United States